CLINICAL TRIAL: NCT01717157
Title: An Open-Label, Randomized, 4-Way Crossover Study to Assess the Relative Bioavailability of 4 New Formulations of Fentanyl Transdermal System Compared Against DUROGESIC Fentanyl Transdermal Patch After Single Application in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability of 4 Formulations of Fentanyl Transdermal System Compared Against DUROGESIC Fentanyl Transdermal Patch After Single Application in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100879; FENPAI1022 (Other: Janssen Research & Development, LLC); 2012-000705-71 (EudraCT Number)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Healthy; Fentanyl; Transdermal patch; DUROGESIC
MeSH Terms: interventions — Fentanyl

ARMS (8):
- Treatment sequence 1 (AEBD) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 2 (BACE) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 3 (CBDA) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl)
- Treatment sequence 4 (EDAC) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 5 (DECA) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 6 (EADB) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 7 (ABEC) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl)
- Treatment sequence 8 (BCAD) (Experimental)
  Interventions: Drug: Treatment A: DUROGESIC (8.4 mg fentanyl); Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl); Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl); Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl)

INTERVENTIONS:
Drug: Treatment A: DUROGESIC (8.4 mg fentanyl) — One DUROGESIC transdermal patch containing 8.4 mg of fentanyl applied on the skin for 72 hours.
Drug: Treatment B: Transdermal System-Concept 1 (6.2 mg fentanyl) — One transdermal system-concept 1 patch containing approximately 6.2 mg of fentanyl applied on the skin for 72 hours.
  Arms: Treatment sequence 1 (AEBD); Treatment sequence 2 (BACE); Treatment sequence 3 (CBDA); Treatment sequence 6 (EADB); Treatment sequence 7 (ABEC); Treatment sequence 8 (BCAD)
Drug: Treatment C: Transdermal System-Concept 2 (6.2 mg fentanyl) — One transdermal system-concept 2 patch containing approximately 6.2 mg of fentanyl applied on the skin for 72 hours.
  Arms: Treatment sequence 2 (BACE); Treatment sequence 3 (CBDA); Treatment sequence 4 (EDAC); Treatment sequence 5 (DECA); Treatment sequence 7 (ABEC); Treatment sequence 8 (BCAD)
Drug: Treatment D: Transdermal System-Concept 3 (7.1 mg fentanyl) — One transdermal system-concept 3 patch containing approximately 7.1 mg of fentanyl applied on the skin for 72 hours.
  Arms: Treatment sequence 1 (AEBD); Treatment sequence 3 (CBDA); Treatment sequence 4 (EDAC); Treatment sequence 5 (DECA); Treatment sequence 6 (EADB); Treatment sequence 8 (BCAD)
Drug: Treatment E: Transdermal System-Concept 4 (11.0 mg fentanyl) — One transdermal system-concept 4 patch containing approximately 11.0 mg of fentanyl applied on the skin for 72 hours.
  Arms: Treatment sequence 1 (AEBD); Treatment sequence 2 (BACE); Treatment sequence 4 (EDAC); Treatment sequence 5 (DECA); Treatment sequence 6 (EADB); Treatment sequence 7 (ABEC)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and relative bioavailability of 4 new formulations of fentanyl transdermal patch in healthy participants after a single application for 72 hours.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study drug is assigned by chance), 4-way crossover (participants will receive different interventions sequentially during the trial) study. The study will assess the pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) and relative bioavailability (the extent to which a drug or other substance becomes available to the body) of 4 new formulations of fentanyl transdermal patch, TDS-Concept 1 50 µg/h, TDS-Concept 2 50 µg/h, TDS-Concept 3 50 µg/h and TDS-Concept 4 100 µg/h compared with DUROGESIC fentanyl 50 µg/h in healthy participants after a single application. All participants will be randomly assigned to 1 of 8 possible treatment sequences. During the 4 single-application treatment periods, each transdermal patch will be worn, on a different application site on the lateral side of the upper arm, continuously for 72 hours. The treatment periods will be separated by a washout period (period when receiving no treatment) of at least 8 and no more than 14 days. The total study length is from 64 days to a maximum of 82 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Participants must utilize a medically acceptable method of contraception throughout the entire study period including the washout period and for 3 months (men) or 1 week (women) after the study is completed
* Men must not donate sperm from the first drug administration until 3 months after completion of the study
* Each participant will receive a test for opioid dependency. Only those participants that pass this challenge test will be allowed to continue in this study
* Non-smoker

Exclusion Criteria:

* History of or current clinically significant medical illness, disease or condition that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Clinically significant abnormal laboratorial values
* Clinically significant abnormal physical examination, vital signs or electrocardiogram (ECG)
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, oral contraceptives and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Fentanyl serum concentrations | Up to 120 hours after applying the transdermal patch
Determination of residual fentanyl content in the worn patchs | At the end of 72 hours after applying the transdermal patch
  The fentanyl content in the patchs following their removal at the end of 72 hours
The skin adherence score of the patches | Up to 72 hours after applying the transdermal patch
  The patch adherence will be scored from 0 to 4, where 0: >= 90% of the area adhered and no edges unattached; 1: >= 75% to < 90% adhered; 2: >= 50% and < 75% adhered; 3: > 0% and < 50% adhered, but not detached; 4: 0% adhered - patch detached.

SECONDARY OUTCOMES:
The incidence of adverse events | Approximately 82 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium